CLINICAL TRIAL: NCT06056739
Title: Alio WEAR Study: Long-term Wear of the Alio Platform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AM23
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Alio platform.
  Interventions: Device: Alio platform
- Control Subject (No Intervention): All subjects who are enrolled into the control group and participate in data collection will not receive the noninvasive Alio platform.

INTERVENTIONS:
Device: Alio platform — Remote monitoring platform
  Arms: Test Subject

SUMMARY:
The WEAR study is long-term interventional study designed to evaluate patient and clinician use of the Alio platform, per its FDA cleared indications.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Receiving hemodialysis via an AVF or AVG in an arm location at the time of study start.
* Able to wear the SmartPatch effectively at the specified location on the arm.
* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
* Willing and able to wear the SmartPatch as instructed and comply with all interviews, surveys and questionnaires, and schedule of evaluations.

Exclusion Criteria:

* Skin near the proximity of the AV access that is chronically swollen, infected, inflamed, open wounds, lesions, or has skin eruptions.
* Participation in any other clinical trials involving investigational or marketed products that in the opinion of the investigator could affect the quality of the data.
* Other conditions that in the opinion of the Principal Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessing usage of the Alio platform by the test subject | Up to 1 year
  Assessing compliance and ease of use via surveys

CONTACTS AND LOCATIONS:
Overall Officials: David Whittaker, MD, Study Director — Alio
Locations (1):
- Site 1, Huntley, Illinois, United States